CLINICAL TRIAL: NCT01719172
Title: A Prospective, Multi-Center, Single-Arm Study of the Veriset™ Hemostatic Patch in Controlling Bleeding in Soft Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVEUST0278
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Non-emergent, Soft Tissue Procedures, Performed Via an Open Approach

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Veriset™ Hemostatic Patch (Experimental): Topical hemostat
  Interventions: Device: Veriset™ Hemostatic Patch

INTERVENTIONS:
Device: Veriset™ Hemostatic Patch — Topical Hemostat

SUMMARY:
The objective of this study is to determine the safety of Veriset™ Hemostatic Patch when used during non-emergent, open, soft tissue surgery where a topical hemostatic agent would be used.

ELIGIBILITY:
Inclusion Criteria:

* Subject or authorized representative has provided informed consent.
* Subject is ≥ 18 years old.
* Subject is scheduled for nonemergent surgery where a topical hemostatic agent would be used to control bleeding emanating from a tissue bed following organ dissection or removal or a bleeding tumor tissue bed following resection or dissection, via an open approach.
* Subject is willing and able to comply with all aspects of the treatment and evaluation schedule.
* Subject has an appropriate Target Bleeding Site (TBS) during the surgical procedure.
* TBS bleeding assessment is Type 2 or 3 (refer to table in protocol).

Exclusion Criteria:

* Subject is pregnant (documented by a positive pregnancy test) or is actively breast-feeding.
* Subject has an estimated life expectancy of less than 6 months.
* Subject is scheduled for another planned surgery and the subsequent surgery would jeopardize the previous application of study treatment.
* Subject is undergoing emergency surgery, i.e. lifesaving procedures performed where patient is in imminent danger of death.
* Subject has participated in an investigational drug or device research study within 30 days of enrollment that would interfere with the study.
* Subject has an active local infection at the TBS.
* The investigator determines that participation in the study may jeopardize teh safety or welfare of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Innsbruck, Austria
- Germany (2):
  - Hanover
  - München

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who were scheduled for non-emergent, soft tissue procedures performed via an open approach were assessed for potential study eligibility via a screening/baseline assessment performed within 30 days of their scheduled procedure.
Pre-assignment Details: Subjects who met the pre-operative eligibility criteria were considered for study participation. During the surgical procedures, subjects who met the intra-operative eligibility criteria were enrolled into the study. Subjects who did not meet all criteria were considered screen failures and not enrolled.
Groups:
- Veriset™ Hemostatic Patch: Subjects received the topical hemostat Veriset™ Hemostatic Patch
Period: Overall Study
Arm/Group | Veriset™ Hemostatic Patch
Started | 30
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographic and clinical characteristics are summarized by descriptive statistics for continuous variables, and frequencies and percentages for categorical variables. These analyses were performed on the Treated Population.
Arm/Group | Veriset™ Hemostatic Patch
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: centimeters] | 174.0 (7.6)
Weight [Mean (Standard Deviation); unit: kilograms] | 75.0 (19.0)

OUTCOME MEASURES:

1. Primary Outcome: Percent Success in Obtaining Hemostasis Following Veriset Hemostatic Patch Treatment
Description: Success will be defined as hemostasis obtained within 5 minutes. Hemostasis will be assessed every 30 seconds until the 5-minute time point, at which point the visual inspection will continue at one-minute intervals up to 10 minutes or until hemostasis is achieved.
Time Frame: Intra-operative (Day 0)
Measure: Number; unit: participants
Arm/Group | Veriset™ Hemostatic Patch
Number analyzed (Participants) | 30
participants | 29
Statistical Analysis 1: Comparison: Veriset™ Hemostatic Patch; The primary effectiveness endpoint was the percent (%) success in obtaining hemostasis at the Target Bleeding Site (TBS) within 5 minutes following Veriset™ application. An exact (Clopper-Pearson) 95% confidence interval for the true success percentage was calculated. Subjects who received rescue therapy on the target bleeding site prior to obtaining hemostasis were considered failures; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — The p-value from a one-sided exact test was based on the binomial distribution, testing that the true percent success rate was ≤ 50% versus the alternative hypothesis that the success rate was > 50%

2. Secondary Outcome: Proportion of Subjects Who Achieve Hemostasis Within 1 Minute
Description: Hemostasis will be assessed every 30 seconds until the 5-minute time point, at which point the visual inspection will continue at one-minute intervals up to 10 minutes or until hemostasis is achieved.
Time Frame: Intra-operative (Day 0)
Measure: Number; unit: participants
Arm/Group | Veriset™ Hemostatic Patch
Number analyzed (Participants) | 30
participants | 21 [50.6 to 85.3]
Statistical Analysis 1: Comparison: Veriset™ Hemostatic Patch; The number and percentage of subjects who achieved hemostasis within 1 minute were presented. An exact (Clopper-Pearson) 95% confidence interval for the true percentage was calculated; Test type: Superiority or Other; p = 0.0214, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Median Time to Achieve Hemostasis
Description: as for outcome 2
Time Frame: Intra-operative (Day 0)
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Veriset™ Hemostatic Patch
Number analyzed (Participants) | 30
Minutes | 1 [0.5 to 1.0]
Statistical Analysis 1: Comparison: Veriset™ Hemostatic Patch; Time to achieve hemostasis was analyzed using the Kaplan-Meier method to estimate the survival distribution and to obtain the estimated median time to hemostasis. Additionally, A 95% Brookmeyer-Crowley confidence interval for the median was computed based on the sign test; Test type: Superiority or Other; Median Difference (Final Values) = 1.0, 95% CI 1-sided [upper limit 1.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 90 day follow-up visit.
Description: All adverse events were reported, regardless of relationship to study device.
Arm/Group | Veriset™ Hemostatic Patch
Serious Adverse Events (participants affected / at risk) | 11/30
Other Adverse Events (participants affected / at risk) | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Veriset™ Hemostatic Patch (N=30)
Atrial fibrillation (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1
Mesenteric haemorrhage (Gastrointestinal disorders) | 1
Impaired healing (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Bacterial diarrhoea (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Laboratory test abnormal (Investigations) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Veriset™ Hemostatic Patch (N=30)
Anaemia (Blood and lymphatic system disorders) | 4
Duodenitis (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Impaired healing (General disorders) | 4
Seroma (Injury, poisoning and procedural complications) | 2
Hepatic enzyme increased (Investigations) | 2
Fluid retention (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3
Renal impairment (Renal and urinary disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No